CLINICAL TRIAL: NCT02994914
Title: GEriatric Determinants of Curative RAdiotherapy Scheme Choice for Breast Cancer ELderly Patient Treatment Compliance and Tolerance : GERABEL Study
Brief Title: GEriatric Determinants of Curative RAdiotherapy Scheme Choice for Breast Cancer ELderly Patient Treatment Compliance and Tolerance
Acronym: GERABEL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low rythm of inclusions
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Centre Antoine Lacassagne (Other); Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-0902; 2016-A01469-42 (Other: ANSM)
Record Dates: First submitted 2016-09-21; First posted 2016-12-16 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Onco Geriatric Evaluation; Radiotherapy; Hypo fractionated radiotherapy; Normo fractionated radiotherapy; Large hypo fractionated radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Score of the Onco Geriatric Evaluation between 200 et 160 (Experimental): According to the score obtained with the onco geriatric evaluation, patients with a score between 200 and 160 will receive a normo fractionated radiotherapy (66 Grays in 33 fractions). This scheme of radiotherapy is already used in the clinical practice, but not allocated according to a score obtained at an oncogeriatric evaluation.
  Interventions: Other: Onco Geriatric Evaluation
- Score of the Onco Geriatric Evaluation between 159 et 120 (Experimental): According to the score obtained with the onco geriatric evaluation, patients with a score between 159 and 120 will receive an hypo fractionated radiotherapy (42,56 Grays in 16 fractions). This scheme of radiotherapy is already used in the usual practice, but not allocated according to a score obtained at an oncogeriatric evaluation.
  Interventions: Other: Onco Geriatric Evaluation
- Score of the Onco Geriatric Evaluation inferior to 119 (Experimental): According to the score obtained with the onco geriatric evaluation, patients with a score inferior to 119 will receive a large hypo fractionated radiotherapy (30 Grays in 5 weekly fractions). This scheme of radiotherapy is already used in the usual practice, but not allocated according to a score obtained at an oncogeriatric evaluation.
  Interventions: Other: Onco Geriatric Evaluation

INTERVENTIONS:
Other: Onco Geriatric Evaluation — Seven tests will be performed by an onco geriatrician : Activities of Daily Living, Instrumental Activities Of Daily Living, Mini Mental State Examination, mini Geriatric Depression Scale, Mini Nutritional Assessment, Cumulative Illness Rating Scale-Geriatric, and " timed get up and go " tests. Those tests lead to a score, and this score will determine the scheme of patients radiotherapy.

SUMMARY:
This study proposes an onco geriatric evaluation (Activities of Daily Living, Instrumental Activities Of Daily Living, Mini Mental State Examination, mini Geriatric Depression Scale, Mini Nutritional Assessment, Cumulative Illness Rating Scale-Geriatric, and " timed get up and go " tests) for elderly breast cancer patients. The score obtained at this evaluation will determine the radiotherapy scheme.

DETAILED DESCRIPTION:
Breast cancer is the most frequent cancer for elderly women and represents the first mortality cause for them. Breast cancer incidence increases for elderly women and will become a major public health problem in the next years.

The principal therapeutic solution is the partial mastectomy associated to radiotherapy. However, the radiotherapy scheme and its role are debated for elderly patients. Hypo fractionated radiotherapy could be considered as an advantageous option.

The treatment duration (6,5 weeks) and direct and indirect fatigue (around 33 travels) are major cons. Thereby, for elderly patients, the selection of patients who will benefit from a shorter treatment could be really difficult. It would be interesting to define an objective scoring, predicting a bad or good tolerance and observance to the radiotherapy. Nowadays, onco geriatric evaluations are used to decide some treatment's decision, but no study compared different orientated radiotherapy schemes.

The present study proposes an onco geriatric evaluation leading to a score according to seven tests (Activities of Daily Living, Instrumental Activities Of Daily Living, Mini Mental State Examination, mini Geriatric Depression Scale, Mini Nutritional Assessment, Cumulative Illness Rating Scale-Geriatric, and " timed get up and go " tests). The score will then determine an adapted radiotherapy scheme.

ELIGIBILITY:
Inclusion Criteria:

* Woman more than 70 years old,
* Patient carrying a breast cancer proven histologically and treated by radiotherapy in curative intent.

Exclusion Criteria:

* Man,
* Patient with metastatic cancer,
* Patient with impossible follow-up at 6 months (planned relocation, patient support in another Center),
* Patient under protection of justice or unable to give consent.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Measure of the tolerance | Month 6
  Tolerance is considered as " bad " if the score of the onco geriatric evaluation decreases of more than 20% from the initial evaluation to 6 months after the end of the rays. Tolerance is considered as "correct" in the other cases.

SECONDARY OUTCOMES:
Tolerance | Month 6
  Specific tolerance will be evaluated by the number of radiation-induced toxicities (Common Terminology Criteria for Adverse Events 4.4) of I, II, III, and IV grades.
Quality of Life Questionnaire | Month 6
  Quality of life will be assessed with the difference between the Quality of Life Questionnaire 30 of the European Organisation for Research and Treatment of Cancer (EORTC) score obtained before the radiotherapy and 6 months after the end of the radiation therapy.
Radiotherapy compliance | Month 6
  Compliance is considered as "bad" if the treatment plan is interrupted for at least one day (for medical reason). Compliance is considered as "correct" in the other cases.
Correlation between tolerance and distance from the therapeutic center | Month 6
  Correlation will potentially be established between patient general tolerance and the distance between home and radio therapeutic center.
Correlation between tolerance and way of transport | Month 6
  Correlation will potentially be established between patient general tolerance and the way of transport used by the patient to go to the therapeutic center.
Correlation between tolerance and the number of concomitant treatments | Month 6
  Correlation will potentially be established between patient general tolerance and the number of concomitant treatments.
Correlation between tolerance and the nature of concomitant treatments | Month 6
  Correlation will potentially be established between patient general tolerance and the nature of concomitant treatments.
Correlation between tolerance and the supportive cares | Month 6
  Correlation will potentially be established between patient general tolerance and the supportive cares performed.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Magné, PhD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (3):
- France (3):
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Groupement Hospitalier Portes de Provence, Montélimar
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No